CLINICAL TRIAL: NCT02733224
Title: Adherence to Lenalidomide Treatment in Multiple Myeloma - Prevalence, Characteristics and Clinical Significance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Irina Amitai, Dr, Rabin Medical Center
Other Study IDs: 0336-15
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Patient Non-adherence
Keywords: lenalidomide adherence MEMS
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
we intend to evaluate the association between non-adherence to Lenalidomide in Multiple Myeloma (MM) patients and overall response rates and time to progression (TTP).

Adherence will be measured in several ways, including by electronic monitoring, which is the gold standard method.

DETAILED DESCRIPTION:
Study Hypothesis: We hypothesize that non-adherence to lenalidomide in MM patients is associated with decreased overall response rates and shorter time to progression (TTP).

Study Objectives:

Primary Objective: To evaluate the association between non-adherence to lenalidomide in MM patients and the overall response rate at 6 months.

Secondary Objectives: 1) To evaluate the prevalence of non-adherence to lenalidomide in MM patients, and independent risk factors thereof. 2) To validate the utility of questionnaires assessing adherence in identifying MM patients at risk for lenalidomide non-adherence.3) To assess the association between non-adherence to lenalidomide and long-term response, measured as time to progression (TTP) at 18 months.

Background: Lenalidomide-based regimens are a key component of the armamentarium for initial treatment in newly diagnosed multiple myeloma patients. Real-life data shows CR rates that are comparable to or slightly higher 1than those seen in prospective clinical trials. This variable response is a result of differences in clinical settings and patient and disease characteristics, but in theory, also may be due to variable adherence to lenalidomide. The development of oral anticancer therapies, such as lenalidomide, represents a significant step forward in oncology care by providing patients with convenient treatment of proven clinical efficacy, but also presents healthcare professionals with the challenge of monitoring and maintaining patients' adherence to this therapy.

Non-adherence may be defined, for example, as non-perfect adherence (i.e. less than 100%), another cutoff with proven clinical significance, or simply as a numerical value representing the percentage of medication taken, relative to that recommended. This definition, together with the method used to measure adherence, can greatly influence reported rates of non-adherence in any given clinical setting. Taking all these limitations into account, reported rates of non-adherence to oral anti-cancer regimens across empirical studies average approximately 25% 2,3.Accordingly, using pharmacy refill data, a recent retrospective study demonstrated that 33% of newly diagnosed MM patients were non-adherent to lenalidomide treatment (defined as adherence < 80%)4. This is the only study, assessing adherence to lenalidomide in MM patients, which we are aware of.

Using electronic monitoring (EM), Marin et al prospectively demonstrated that poor adherence to the tyrosine kinase inhibitor (TKI), imatinib, in CML, adversely impacts molecular and cytogenetic response 5,6.This landmark study provided proof of concept that non-adherence to oral anti-cancer in hematological malignancies may be associated with poor responses and decreased survival. Our study group is currently analyzing data from our prospective interventional study aimed at improving adherence to TKIs in CML (NCT01768689).

In light of this evidence, in an era that has witnessed the advent of effective oral agents for MM, understanding the prevalence, characteristics and clinical implications of non-adherence to these agents is key to providing high-quality care for these patients. Nevertheless, research regarding adherence to oral agents in MM (e.g. thalidomide, lenalidomide, pomalidomide) is still in its infancy, and there are no data indicating whether a similar association between adherence and treatment response exists in this field. Moreover, there is a paucity of data regarding the prevalence of non-adherence and risk factors thereof, in the above context.

Study design:

Prospective multi-center observational (non-interventional) cohort study.Patients will be managed routinely according to the local protocol at each center for the treatment of multiple myeloma. Study period: From initiation of lenalidomide therapy for a period of 18 months. Setting and location: Institute of hematology, Sheba medical center and Hematology Institute at the Davidoff cancer center, Rabin medical center, Israel.

Inclusion criteria: Patients diagnosed with active MM starting induction treatment with the lenalidomide with or without dexamethasone, as any line of therapy.

Key exclusion criteria: Treatment with any additional anti-myeloma drugs, during study period.

Patient characteristics and confounders: Patient characteristics (demographics, comorbidities); Disease-related characteristics (duration, myeloma stage and risk, details regarding previous therapy and response, functional status, quality of life); Other drugs (Number of drugs, pills and potential interactions with lenalidomide). We will use an adaptation of the questionnaire from the "BRIGHT" study (which assesses barriers to immunosuppressive medication adherence in heart transplant recipients) to assess barriers to adherence in this patient cohort.

Measurement of adherence: Adherence to lenalidomide treatment will be measured continuously throughout the study period, by several means: 1) Electronic monitoring (EM) will be used throughout the first 5 months of the study period. This is considered the gold standard for measuring adherence, reflecting adherence more objectively than questionnaires and pill-counting. The microelectronic monitoring system (MEMS), a specific type of EM, consists of an electronic device ﬁtted in the cap of a normal-looking medication bottle that automatically records each time the bottle is opened. Adherence measured with this device was associated with treatment response in the landmark study in CML by Marin et al. 2) Pill counting for first five months. 3) Questionnaires: The physician visual analogue scale (physician VAS) and an adaptation of the "Basel assessment of adherence with the Immunosuppressive Regimen Scale" (BAASIS), will be assessed at predefined time points throughout the 18 months of the study period.

Outcome Measures: Primary outcome measure: Response to treatment (Overall response) 4 weeks after finishing five months of electronic adherence monitoring (i.e. at 6 months).

Analysis: Primary analysis: Incidence of the primary outcome measure in patients with electronically measured adherence of above 90% versus those below 90%, as measured for 5 consecutive months after study initiation.

Secondary analysis: 1) Analyze the association of each of the baseline characteristics / confounders and adherence-barriers questionnaire to electronically-measured adherence and look for independent risk factors for non-adherence. This will be stratified to line of treatment. 2) Validation of study questionnaires compared to electronically measured adherence.

3) A long-term analysis which will look at an association between TTP at 18 months and both initial adherence measure electronically (first 5 months) and long term overall adherence measured by BAASIS questionnaire (18months).

Sample size:

In a prior study7, the ORR (i.e. PR and better) was 68% in the Rd arm, after 4 cycles. A prior study in CML showed a profound effect of adherence above 90% on optimal treatment response (RR=11) 5. As no data exists regarding the effect of adherence on outcome in our study population we utilized a RR which was conservative (<2), relative to the data from CML. We assumed an 80% ORR at 6 months in the adherent group and 45% ORR at 6 months in the non-adherent group (defined by a cutoff of 90% adherence). Prior data8 suggested the adherent/non-adherent ratio in patients receiving lenalidomide induction for myeloma is 7:3, and we assumed a similar ratio of 2:1.

Based on the above data, we calculated that 43 patients in the adherent arm and 22 patients in the non-adherent arm will have a power of 0.8 (with a type I error of 0.05) to reject the null hypothesis that there is no difference in ORR between these groups.

Therefore the required sample size is 67.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with active MM
* starting induction treatment with lenalidomide with or without dexamethasone
* any line of therapy.

Exclusion Criteria:

* Treatment with any additional anti-myeloma drugs, during study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with active MM starting induction treatment with the lenalidomide with or without dexamethasone, as any line of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Response to treatment (Overall response) 4 weeks after finishing five months of electronic adherence monitoring (i.e. at 6 months). | within 4 weeks after 5 months of follow-up

IPD SHARING:
Plan to Share IPD: No